CLINICAL TRIAL: NCT07385534
Title: Effects of Lower Body Electrical Muscle Stimulation Training on Body Composition, Muscle Function, and Arteriosclerosis Markers in Postmenopausal Women
Brief Title: Effects of Lower Body EMS Training in Postmenopausal Women
Acronym: LB-EMS-PMW
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University (Other)
Responsible Party: Principal Investigator, Kyungho Kim, Principal Investigator, Seoul National University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB No. 2601/002-017
Record Dates: First submitted 2026-01-23; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Sarcopenia; Arteriosclerosis; Arterial Stiffness, Blood Pressure; Postmenopausal Women
Keywords: Electrical Muscle Stimulation; EMS; Resistance Training; Postmenopausal Women; Body Composition; Vascular Health; Muscle Function
MeSH Terms: conditions — Sarcopenia; Arteriosclerosis

STUDY DESIGN:
Intervention Model Description: A parallel-group design with three arms: 1) Lower Body EMS combined with Resistance Training, 2) Resistance Training alone, and 3) Control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lower Body EMS + Resistance Training Group (Experimental): Participants perform lower body resistance training while wearing a lower body EMS suit. Each session lasts 50 minutes (10-min warm-up, 30-min main exercise, 10-min cool-down). EMS stimulation is applied exclusively during the 30-minute main exercise phase (85Hz, 350µs). This program is conducted twice a week for 6 weeks.
  Interventions: Device: Lower-body Electromyostimulation (LB-EMS) device; Behavioral: Lower Body Resistance Training
- Resistance Training Only Group (Active Comparator): Participants perform the identical lower body resistance training program without EMS stimulation. The session structure (10-min warm-up, 30-min main exercise, 10-min cool-down) and total duration (50 minutes) are the same as the experimental group.
  Interventions: Behavioral: Lower Body Resistance Training
- Control Group (No Intervention): Participants maintain their usual daily lifestyle without engaging in any new exercise programs during the 6-week study period.

INTERVENTIONS:
Device: Lower-body Electromyostimulation (LB-EMS) device — Electrical stimulation applied to the lower body muscles (85Hz, 350µs) during the main exercise phase
  Arms: Lower Body EMS + Resistance Training Group
Behavioral: Lower Body Resistance Training — A 50-minute session consisting of a 10-minute warm-up, 30 minutes of main lower body resistance training (4 types of machine-based exercises per session), and a 10-minute cool-down
  Arms: Lower Body EMS + Resistance Training Group; Resistance Training Only Group

SUMMARY:
This study evaluates the effects of a 6-week lower body Electrical Muscle Stimulation (EMS) training program on body composition, muscle function, and arteriosclerosis markers in postmenopausal women.

Menopause is associated with a rapid decline in estrogen, which increases the risk of sarcopenia (muscle loss) and arterial stiffness (cardiovascular disease). While resistance training is effective for these conditions, participation rates among postmenopausal women are often low. This study investigates whether applying EMS during lower body resistance exercises provides superior benefits compared to resistance training alone or no intervention.

Participants will be randomized into three groups:

1. Lower-body EMS combined with Resistance Training Group
2. Resistance Training Only Group
3. Control Group (No intervention)

The study aims to verify the efficacy of EMS as a time-efficient and effective alternative exercise modality for improving vascular and musculoskeletal health in this population.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women (defined as cessation of menstruation for at least 12 months).
* Aged between 50 and 70 years.
* Sedentary lifestyle (no participation in regular resistance training programs within the last 6 months).
* Able to perform lower body resistance exercise with LB-EMS suit.
* Willing to participate in the study and provide informed consent.

Exclusion Criteria:

* Contraindications for WB-EMS: Presence of implanted electrical devices (e.g., pacemakers, defibrillators), severe bleeding disorders (e.g., hemophilia), abdominal/inguinal hernia, or history of surgery within the last 6 months (including stent insertion).
* Severe Chronic Diseases: Diagnosis of severe cardiovascular (e.g., MI, heart failure, arrhythmia), renal, neurological (e.g., epilepsy), or oncological diseases (currently undergoing treatment).
* Uncontrolled Cardiovascular Conditions: Uncontrolled hypertension or severe arterial circulatory disorders.
* Confounding Medications: Current use of hormone replacement therapy (HRT) for menopause or medications for severe psychiatric disorders (e.g., depression, anxiety).
* Acute Conditions & Others: Acute infection/inflammation, influence of alcohol/drugs, or any other condition deemed unsuitable by the investigator.

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2025-12-26 (Actual); Primary Completion 2026-03-26 (Estimated); Study Completion 2026-05-26 (Estimated)

PRIMARY OUTCOMES:
Brachial-ankle Pulse Wave Velocity (baPWV) | Baseline and Week 6
  An indicator of arterial stiffness. Higher values indicate stiffer arteries. Unit of Measure: cm/s

SECONDARY OUTCOMES:
Ankle-Brachial Index (ABI) | Baseline and Week 6
  The Ankle-Brachial Index (ABI) is the ratio of the systolic blood pressure measured at the ankle to the systolic blood pressure measured at the brachial artery. It is a non-invasive indicator used to assess the presence and severity of peripheral arterial stenosis or occlusion. Lower ABI values (typically < 0.9) suggest narrowing or blockage of the arteries in the legs.
  Unit of Measure: ratio
Skeletal Muscle Mass | Baseline and Week 6
  Assessed using Bioelectrical Impedance Analysis (BIA). Represents the total weight of muscle tissue attached to the skeleton. Unit of Measure: kg
Total Body Fat Mass | Baseline and Week 6
  Assessed using BIA. Represents the total weight of adipose tissue in the body. Unit of Measure: kg
Body Fat Percentage | Baseline and Week 6
  Assessed using BIA. The proportion of fat mass relative to total body weight. Unit of Measure: %
Extracellular Water to Total Body Water Ratio (ECW/TBW) | Baseline and Week 6
  Assessed using BIA. An indicator of body fluid balance and edema. Higher values may indicate fluid retention or inflammation.
  Unit of Measure: ratio
Skeletal Muscle Mass Index (SMI) | Baseline and Week 6
  Calculated as appendicular skeletal muscle mass (ASM) divided by height squared (kg/m^2). Used to assess sarcopenia status.
  Unit of Measure: kg/m^2
Phase Angle | Baseline and Week 6
  Assessed by BIA. It reflects cellular membrane integrity and nutritional status. Higher values generally indicate better cellular health.
  Unit of Measure: degree
Pre-ejection Period (PEP) | Baseline and Week 6
  Time interval from the onset of ventricular depolarization (QRS complex) to the beginning of ejection. Reflects myocardial contractility. Unit of Measure: ms
Left Ventricular Ejection Time (ET) | Baseline and Week 6
  The duration of blood flow ejection from the left ventricle into the aorta. Unit of Measure: ms
Heart Rate Corrected Ejection Time (ETc) | Baseline and Week 6
  Ejection time adjusted for heart rate, typically using Bazett's formula. Unit of Measure: ms
Upstroke Time (UT) | Baseline and Week 6
  Time from the foot to the peak of the pulse volume waveform. A marker for arterial stiffness or stenosis.
  Unit of Measure: ms
ET/PEP Ratio | Baseline and Week 6
  The ratio of ejection time (ET) to pre-ejection period (PEP). An index of left ventricular performance and efficiency.
  Unit of Measure: ratio
Percent Mean Arterial Pressure (%MAP) | Baseline and Week 6
  The position of mean arterial pressure relative to the pulse pressure range. Used as an indicator of the pulse wave shape and vascular aging.
  Unit of Measure: %
Mean Arterial Pressure (MAP) | Baseline and Week 6
  The average pressure in a patient's arteries during one cardiac cycle. Unit of Measure: mmHg
Pulse Pressure (PP) | Baseline and Week 6
  The difference between systolic and diastolic blood pressure. It is a marker of arterial stiffness.
  Unit of Measure: mmHg
Peak Torque (Knee Extension/Flexion) | Baseline and Week 6
  The maximum torque produced during isokinetic knee extension and flexion. Assessed at a 60°/s angular velocity.
  Unit of Measure: Nm (Newton-meters)
Total Work Done | Baseline and Week 6
  The total amount of work performed by the muscle groups during the test protocol at an angular velocity of 180°/s.
  Unit of Measure: Nm
Fatigue Index | Baseline and Week 6
  The percentage decline in peak torque calculated from the difference between the initial and final repetitions during a set of isokinetic contractions performed at an angular velocity of 180°/s.
  Unit of Measure: %
Hamstring-Quadriceps Ratio (H/Q Ratio) | Baseline and Week 6
  The ratio of the peak torque of the hamstring muscles to the peak torque of the quadriceps muscles measured at an angular velocity of 60°/s.
  Unit of Measure: ratio
Bilateral Deficit | Baseline and Week 6
  The percentage difference between the sum of peak torques produced by each leg individually and the peak torque produced when both legs act simultaneously, measured at an angular velocity of 60°/s.
  Unit of Measure: %

CONTACTS AND LOCATIONS:
Overall Officials: Yeon Soo Kim, MD, Principal Investigator — Seoul National University
Locations (1):
- Seoul National University, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No